CLINICAL TRIAL: NCT00262496
Title: Botulinum-A Toxin Injection for Detrusor Hyperreflexia in Spinal Cord Injury: A Non-Surgical Approach.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3216-01
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Overactive Bladder; Urinary Incontinence
Keywords: Botox; Overactive bladder; Incontinence; Spinal Cord Injury
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence; Spinal Cord Injuries | interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: Botox

SUMMARY:
The purpose of the study is to determine whether Botulinum-A toxin injected in the bladder muscle will help prevent the frequency and degree of urinary incontinence in Spinal Cord Injured and Multiple Sclerosis patients. The proposed mechanism would be that the Toxin would allow the bladder to hold more urine at a lower pressure as determined by Urodynamics. The research will answer the question whether the dosages 300 units vs 400 units are either equally vs not equally effective in helping urinary incontinece and bladder storage.

DETAILED DESCRIPTION:
OBJECTIVE OF THE PROJECT The major aim of the present study is to use a double blind randomized clinical trial design to evaluate the long-term efficacy and safety of two different doses, 300 and 400 Units of Botulinum Toxin Type-A for the treatment of detrusor hyperreflexia (Neurogenic Bladder Overactivity). While also improving bladder capacity in spinal cord injured patients with refractory symptoms who have failed anticholinergic agents.

RESEARCH PLAN Inclusion Criteria: Male and female subjects 18-80 years of age with suprasacral SCI refractory NBOA incontinence, and/or impaired detrusor compliance associated with a small bladder capacity will be eligible. Subjects will be recruited on the basis of incontinence symptoms and adverse urodynamic parameters including impaired bladder compliance less than 50ml/cm, H20 and bladder (cystometric) capacity less than 300 ml.

Exclusion criteria: Allergy to Botulinum Toxin Type-A, pregnancy, breast-feeding women, active medical or psychiatric disorders, active urinary tract infection, coagulopathy, myasthenia gravis, upper urinary tract changes unrelated to lower tract dysfunction, and aminoglycoside use during the last three months. Furthermore, subjects with radiation cystitis (by history), vesico-ureteral reflux (by videofluoroscopy), bladder calculi (by cystoscopy) will be excluded.

Evaluation will include history and physical examination, urine analysis, urine culture and sensitivity, 24-hour voiding diary for 3 consecutive days, urine pregnancy test in female subjects of reproductive age, validated questionnaires, multichannel videourodynamics (UDS), post-void residual volume at the time of UDS, and renal ultrasound.

METHODOLOGY One week after the pre-intervention evaluation, endoscopic injection of Botulinum Toxin Type-A (300 Units or 400 Units) into the detrusor muscle will be performed. During the 24 month duration of the study, participants will take and record their regular bladder medications as Dr. Gousse (or one of his assistants) decide necessary to control their urinary symptoms. Subjects will be scheduled to return at 2, 6, and 12 weeks after the first injection session, and every 3 months thereafter. At the 2-week visit we will assess untoward effects. At the 6-week visit and every subsequent visit a focused physical examination will be carried out, along with validated questionnaires.

Participants with initial success, as defined by 50% improvement (voiding diary) in diminished leakage, improved cystometric capacity by greater than 100 ml, improved compliance by 15 ml/cm H20, 50% improvement in questionnaire scores, but who lose the initial therapeutic benefit will be considered candidates for re-injection every 6 months. Patients who continue to maintain therapeutic benefit pass 6 months after initial injection will not be re-injected and will be re-evaluated at every 3 months thereafter prior to possible re-injection. Pregnancy testing will be obtained prior to each injection session in appropriate female subjects in their reproductive years.

Depending on the type of variable being analyzed different statistical techniques will be used for these comparisons including paired sample t-tests, Wilcoxon's signed rank tests, McNemar's tests, and Cochran's Q tests. Cross-sectional as well as longitudinal analyses will be performed to compare 300 vs. 400 Unit groups with respect to each of the variables ascertained at each time point, and also with respect to changes over time for the major study end points.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18-80 years old with suprasacral spinal cord injury (SCI) or multiple sclerosis (MS) refractory Neurogenic bladder overactivity and/or detrusor compliance associated with small bladder capacity.· Impaired bladder compliance less than 50 ml/cm, H2O and bladder (cystometric) capacity less than 300ml.-

Exclusion Criteria:

* Allergy to Botulinum Toxin Type-A· Pregnancy· Breast-feeding women· Active medical or psychiatric disorders· Upper urinary tract changes unrelated to lower tract dysfunction· Aminoglycoside use during the last 3 months-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angelo E Gousse, MD, Principal Investigator — Miami VA Medical Center
Locations (1):
- Miami VA Medical Center, Miami, Florida, United States

REFERENCES:
- [Background] Schulte-Baukloh H, Weiss C, Schobert J, Stolze T, Sturzebecher B, Knispel HH. [Subjective patient satisfaction after injection of botulinum-a toxin in detrusor overactivity]. Aktuelle Urol. 2005 Jun;36(3):230-3. doi: 10.1055/s-2004-830203. German. PMID 16001338
- [Background] Schurch B, de Seze M, Denys P, Chartier-Kastler E, Haab F, Everaert K, Plante P, Perrouin-Verbe B, Kumar C, Fraczek S, Brin MF; Botox Detrusor Hyperreflexia Study Team. Botulinum toxin type a is a safe and effective treatment for neurogenic urinary incontinence: results of a single treatment, randomized, placebo controlled 6-month study. J Urol. 2005 Jul;174(1):196-200. doi: 10.1097/01.ju.0000162035.73977.1c. PMID 15947626
- [Background] Werner M, Schmid DM, Schussler B. Efficacy of botulinum-A toxin in the treatment of detrusor overactivity incontinence: a prospective nonrandomized study. Am J Obstet Gynecol. 2005 May;192(5):1735-40. doi: 10.1016/j.ajog.2004.11.052. PMID 15902187
- [Background] Bagi P, Biering-Sorensen F. Botulinum toxin A for treatment of neurogenic detrusor overactivity and incontinence in patients with spinal cord lesions. Scand J Urol Nephrol. 2004;38(6):495-8. doi: 10.1080/00365590410015867. PMID 15841785
- [Background] Grosse J, Kramer G, Stohrer M. Success of repeat detrusor injections of botulinum a toxin in patients with severe neurogenic detrusor overactivity and incontinence. Eur Urol. 2005 May;47(5):653-9. doi: 10.1016/j.eururo.2004.11.009. Epub 2005 Jan 15. PMID 15826758
- See also: South Florida VA Foundation for Research — http://sfvafre.org
- See also: American Spinal Injury Association — http://www.asia-spinalinjury.org